CLINICAL TRIAL: NCT00339651
Title: Preliminary Study of Endometrial Hyperplasia: Groundwork for a Study to Define an Optimal Classification of Endometrial Carcinoma Precursors
Brief Title: Preliminary Study of Endometrial Hyperplasia Groundwork for a Study to Define Precursors of Endometrial Cancer
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999903053; 03-C-N053
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Endometrial Hyperplasia; Endometrial Cancer; Postmenopausal Bleeding; Vaginal Bleeding
Keywords: Precursors; Endometrial Cancer; Hyperplasia; Progression
MeSH Terms: conditions — Endometrial Hyperplasia; Endometrial Neoplasms; Uterine Hemorrhage; Hyperplasia; Disease Progression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tissue

GROUPS / COHORTS (2):
- Cases: Women in one large U.S. health care plan. Cases will consist of women who developed endometrial carcinoma or censored complex atypical hyperplasia at least 1 year after receiving a diagnosis of endometrial hyperplasia.
- Controls: Women in one large U.S. health care plan. Controls will consist of individually matched women who received a diagnosis of endometrial hyperplasia at the same age and date as the cases and were cancer-free and hysterectomy-free until the date at which the index cases were diagnosed with endometrial carcinoma or censored complex atypical hyperplasia.

SUMMARY:
This study, conducted jointly by the National Cancer Institute and the Kaiser Permanente Center for Health Research Northwest (KPCHRN) in Portland, Oregon, will lay the groundwork for a future study to identify precursors of endometrial cancer; that is, conditions that precede development of cancer of the lining of the uterus. The diagnosis of endometrial hyperplasia (a condition of abnormal proliferation of endometrial tissue) includes most precursors of endometrial cancer, as well as many benign conditions. Currently, three methods of classifying endometrial cancer precursors have been suggested based on endometrial hyperplasia findings, but it is not known which classification best predicts cancer risk.

This study will examine surgical specimens of hyperplasia and cancer from women diagnosed with endometrial cancer at least 2 years after a diagnosis of endometrial hyperplasia. Investigators will estimate the percentage of cases with different degrees of hyperplasia, and assess the subsequent cancers that developed. This will allow them to rank hyperplasia lesions according to cancer risk and identify lesions that represent the most immediate cancer precursors. They will also review patients medical charts for information related to cancer risk and treatment.

Study participants will include women enrolled in the KPCHRN who are 40 years of age or older and who were diagnosed with endometrial cancer at least 2 years after being diagnosed with endometrial hyperplasia.

DETAILED DESCRIPTION:
Three systems have been proposed to classify endometrial carcinoma precursors, but it is currently unclear which system best predicts cancer risk and is most reproducible. The optimal surrogate endpoint for endometrial carcinoma is therefore unknown. The pathologic diagnosis of endometrial hyperplasia (EH) includes most suspected immediate precursors and many mild, highly reversible proliferations. We propose an exploratory study to assess the feasibility of investigating EH as a source of an endometrial carcinoma surrogate endpoint.

We are conducting a nested case-control study within a large, population-based health care plan. We will identify cases, defined as women who were diagnosed with EH at least one year before being diagnosed with endometrial carcinoma or severe atypical hyperplasia at hysterectomy, through a computerized search of plan databases. We will retrieve the slides from the matching biopsy and hysterectomy on which carcinoma was diagnosed. Women ages 40 or older who were plan members and received a biopsy or curettage diagnosis of EH between 1970 and 2002 will be eligible to be a case.

We will perform an initial histologic review of cases index biopsy slides to assess two types of misclassification known to affect the diagnosis of EH: a) false-negative endometrial carcinoma (i.e., prevalent carcinoma t the time of EH diagnosis) and b) false-positive EH (i.e., a benign, non-hyperplastic lesion). From cases physical records and linked computer records, we will collect data on histopathologic classification of EH lesions and subsequent carcinomas; descriptive data (e.g., patient weight, parity, and menopausal status); and a summary of relevant treatments and follow-up procedures (e.g., hormone therapy or additional clinical procedures).

We will select controls, defined as women who were diagnosed with EH but then did not develop endometrial carcinoma or undergo hysterectomy for a follow-up interval that is equivalent to the follow-up interval of the cases. Controls will be individually matched to cases on age at EH diagnosis, date of EH diagnosis, and duration of follow-up, and also counter-matched based on the original EH diagnosis. After selecting 3 controls per case, we will assemble the same data from controls: histologic review of original slides, descriptive data from medical records databases, and treatment and follow-up procedure data from linked databases.

These data will then be used to estimate the cancer risk associated with specific EH classifications, identify other patient or clinical factors that might modify those risks, explore predictors of EH, and explore molecular factors that might influence the probability of developing carcinoma after a diagnosis of EH.

ELIGIBILITY:
* INCLUSION CRITERIA:

All women who were members of the KPNW health plan between 1970 and 2003 who were at risk of developing endometrial carcinoma will be eligible.

EXCLUSION CRITERIA:

Women will be considered ineligible if they had substantial gaps in KPNW coverage during the years between the index biopsy and diagnosis date (cases) or censoring date (controls).

NCI and KPNW will review otherwise eligible women who have coverage gaps to identify substantial gaps and determine eligibility on an individual basis.

Ages: 40 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We are conducting a nested case-control study of adenocarcinoma of the endometrium within a retrospective cohort of one large managed health care organization in the Northwest U.S. Cases, i.e., women who developed endometrial cancer after a diagnosis of endometrial hyperplasia, will be compared with women who were diagnosed with endometrial hyperplasia but did not develop cancer during an equivalent follow-up period, after controlling for relevant confounders.@@@@@@
Sampling Method: Non-Probability Sample
Enrollment: 745 (Actual)
Dates: Start 2002-11-25 (Actual); Primary Completion 2020-08-06 (Actual); Study Completion 2020-08-06 (Actual)

PRIMARY OUTCOMES:
Endometrial cancer and endometrial hyperplasia. | Cases were diagnosed between 2003 and 2012. Tissue collection is ongoing
  Formalin fixed paraffin embedded tissue blocks and pathology slides from women with endometrial cancer and women with endometrial hyperplasia with covariate data from medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Wentzensen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Kaiser Permanente Northwest, Hillsboro, Oregon, United States

REFERENCES:
- [Background] Skov BG, Broholm H, Engel U, Franzmann MB, Nielsen AL, Lauritzen AF, Skov T. Comparison of the reproducibility of the WHO classifications of 1975 and 1994 of endometrial hyperplasia. Int J Gynecol Pathol. 1997 Jan;16(1):33-7. doi: 10.1097/00004347-199701000-00006. PMID 8986530
- [Background] Bergeron C, Nogales FF, Masseroli M, Abeler V, Duvillard P, Muller-Holzner E, Pickartz H, Wells M. A multicentric European study testing the reproducibility of the WHO classification of endometrial hyperplasia with a proposal of a simplified working classification for biopsy and curettage specimens. Am J Surg Pathol. 1999 Sep;23(9):1102-8. doi: 10.1097/00000478-199909000-00014. PMID 10478671
- [Background] Baak JP, Orbo A, van Diest PJ, Jiwa M, de Bruin P, Broeckaert M, Snijders W, Boodt PJ, Fons G, Burger C, Verheijen RH, Houben PW, The HS, Kenemans P. Prospective multicenter evaluation of the morphometric D-score for prediction of the outcome of endometrial hyperplasias. Am J Surg Pathol. 2001 Jul;25(7):930-5. doi: 10.1097/00000478-200107000-00012. PMID 11420465